CLINICAL TRIAL: NCT01948323
Title: Pregnancy-Related Obesity Prevention Through Education & Communication Technology in AFRICA:The PROTECT-AFRICA STUDY
Acronym: PROTECT-AFRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Prof. Karen Sliwa, Professor, University of Cape Town
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROTAF1402013
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
Keywords: Pregnancy; Maternal health; Newborn health; Information technology; Health education; Cellphone; Touch screen technology; Pregnancy outcome; Low-Middle income; Nurse-led; Nutrition; Exercise
MeSH Terms: conditions — Obesity; Health Education; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- .HEDUAfrica IT package+ std care info (Other): The HEDUAfrica IT package website aims to target disadvantaged gravid women representing the core aspect of the intervention. The website is available on a touch screen panel at the two intervention clinics, (Cape Town and Soweto, SA). A healthcare worker will assist women with the touchscreen tablet at the follow up sessions. The website content includes a number of short videos and health messages related to a pregnancy-specific-disease outcomes. Patients participating in the IT package also receive std car info
  Participants are also asked to complete 2 questionnaires (24 hour dietary recall assessment and short messaging service technology driven) in conjunction to engaging with the HEDUAfrica website. The intervention is standardized across all participants in the intervention group.
  Interventions: Behavioral: HEDUAfrica IT package+ standard care
- Health awareness brochure + std care (No Intervention): Participants in the non-intervention group at another clinic in Soweto, will receive an enhanced form of standard care. This will include, in conjunction with the normal form of care at each clinic,a health awareness brochure that will focus specifically on health information relating to obesity, diabetes, diet, exercise and breastfeeding at each follow-up sessions. These participants will also be asked to fill out the 24 hour dietary recall assessment and short messaging service technology questionnaire (exactly the same as the intervention group) with help from a healthcare worker.

INTERVENTIONS:
Behavioral: HEDUAfrica IT package+ standard care — The HEDUAfrica website aims to target disadvantaged pregnant women representing the core aspect of the intervention. The website is available on a touch screen panel at the two intervention clinics, (Cape Town and Soweto, South Africa). A trained healthcare worker will assist women by means of a touchscreen tablet at the follow up sessions. The website content includes a number of short videos and health messages related to a pregnancy-specific-disease outcomes.
  Participants are also asked to complete 2 questionnaires (24 hour dietary recall assessment and short messaging service technology driven) in conjunction to engaging with the HEDUAfrica website. The intervention is standardized across all participants in the intervention group.
  Arms: .HEDUAfrica IT package+ std care info

SUMMARY:
The purpose of this study is to investigate whether overweight but not obese pregnant African women having unlimited access to a health education-information technology (IT) based intervention package gain weight within the acceptable range of 8-12 kg during the pregnancy period.

Therefore, we hypothesize that unlimited access to health education via an IT-based intervention package has the potential to reduce the onset of obesity in African pregnant women.

To date (Aug 2015), 95% of patients have been recruited, 1320 potential subjects have been screened and 150 enrolled into the study

ELIGIBILITY:
Inclusion Criteria:

* body-mass index (BMI) range of 25.1-29.9 kg/m2
* Weeks of pregnancy: 16-20
* singleton pregnancy

Exclusion Criteria:

* Evidence of pre-existing cardiovascular disease or a metabolic disorder (i.e. gestational diabetes)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To determine a clinically significant difference (absolute difference of ≥10%) in the proportion of participants who gain > 12kg throughout study period will be less in the intervention group compared to the the non-intervention group. | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum

SECONDARY OUTCOMES:
Change in plasma Vitamin C levels in both the mother and newborn | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum; newborn: day of delivery, 6 weeks old, 12 weeks old
Change in blood pressure profiles | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum; newborn: day of delivery, 6 weeks old, 12 weeks old
Improved resting heart rate | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum; newborn: day of delivery, 6 weeks old, 12 weeks old
Clinically normal C-reactive protein levels (<1 mg/dL) | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum; newborn: day of delivery, 6 weeks old, 12 weeks old
Apgar score >3 | Newborn: Day of delivery
To determine what women actually know (and how much they understand) about the risk factors during their pregnancy. | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum
  Mobile intervention with text messages provide essential health information and encouragement to patients which may act as an effective strategy in preventing weight gain which will be assessed with a pre and post intervention questionnaire to evaluate whether the texts were understood and deemed beneficial by the patients.
Improved awareness of food choices | Mother: Baseline (16-20 weeks pregnancy), 24 weeks, 32 weeks, 6 weeks postpartum
  A 24 hour recall dietary assessment will be administered to evaluate changes in food choice behaviour.
Cost saving potential of intervention from a societal perspective. | September 2015
Change in body composition (fat percentage, body water percentage, bone mass, muscle mass, bone density and visceral fat) of mother. | Mother: Baseline (12-16 weeks pregnancy), 24 weeks, 32 weeks, day of delivery, 6 weeks & 12 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sliwa, PhD, Principal Investigator — Hatter Institute for Cardiovascular Research in Africa (HICRA), University of Cape Town
Locations (2):
- South Africa (2):
  - Elias Motsoaledi clinic, Johannesburg, Gauteng
  - Senaoane Clinic, Johannesburg, Gauteng

REFERENCES:
- See also: This is the official website for the Hatter Institute for Cardiovascular Research in Africa. — http://african-heart.org
- See also: This is the official website of the Soweto Cardiovascular Research Heart Unit. — http://www.socru.org
- See also: This is the health education website used in the intervention. — http://www.hedu-africa.org